CLINICAL TRIAL: NCT04229732
Title: Trials of Ventilation Assisted Substance Elimination Via the Lung - Ethanol (VASEL - Ethanol)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Thornhill Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CAPCR ID 15-8982.4
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ClearMate Intervention (Experimental): Participants undergo passive isocapnic hyperventilation via the ClearMateTM device and have regular venous blood samples obtained to measure ethanol clearance kinetics.
  Interventions: Device: ClearMateTM
- Supportive Management (No Intervention): Participants receive standard of care, supportive management, for alcohol intoxication, having regular venous blood samples obtained to measure ethanol clearance kinetics.

INTERVENTIONS:
Device: ClearMateTM — Passive isocapnic hyperventilation breathing circuit.
  Arms: ClearMate Intervention

SUMMARY:
This prospective, randomized control trial will use passive, isocapnic hyperventilation, applied via the ClearMateTM device (Thornhill Medical, Inc) versus controls receiving standard of care supportive management for severe alcohol intoxication to assess for enhanced ethanol elimination kinetics.

ELIGIBILITY:
Inclusion Criteria:

* intoxicated requiring admission to an emergency unit

Exclusion Criteria:

* Liver or renal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Genders will be noted and used for separate analysis due to known gender differences in alcohol elimination kinetics.
Enrollment: 40 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Alcohol elimination time constant | 6-24 hours
  From the recorded venous ethanol blood alcohol values, an elimination time constant will be calculated

IPD SHARING:
Plan to Share IPD: Undecided